CLINICAL TRIAL: NCT02134132
Title: Utilization of Umbilical Cord Blood-derived Platelet Gel for Treatment of Diabetic Foot Ulcers,a Randomized Double Blind Clinical Trial
Brief Title: Utilization of Platelet Gel for Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-PVD-003
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2011-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Platelet gel; diabetic foot ulcer; umbilical cord blood
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet rich plasma (Active Comparator): The patients with diabetic foot ulcer who receive PG treatment.
  Interventions: Biological: Platelet Gel
- Placebo (Placebo Comparator): The patients with diabetic foot ulcer who receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Platelet Gel — Application of platelet gel in patients suffering from diabetic foot ulcers.
  Arms: platelet rich plasma
Other: Placebo — The patients with Diabetic foot ulcer who receive placebo instead of PL Gel.
  Arms: Placebo

SUMMARY:
Diabetes is a multiorgan disease and considered a major health problem in different societies. One of the complications the pain particularly in the extremities resulting from a process known as diabetic foot ulcer. The diabetic patients are subjected to many complications because of foot ulcers, many of them like as chronic wound disease or pressure ulcers (bed sore). Routinely used medical measures for diabetic foot ulcers are depended to nursing care and take too long until pain relief. Among many tested materials and works for wound healing such as debridement, tissue oxygenation, and skin transplantation, platelet-derived compounds are allocated the pivotal position between investigators to tissue regeneration and shortening the wound healing process.

Many of platelet components are procured from platelet rich plasma (PRP) from whole blood donation. Furthermore, it requires to an additional purification step to diminish the volume and facilitate handling in some studies. It means that platelet concentrates (PCs) may be obtained leading to more concentrated platelets in lower volume.

Two types of granules in platelet is responsible for storage of many useful and different growth factors: dense or delta and alpha granules. Platelet-derived growth factors have the ability to growth and differentiation of numerous cells. Also, the antibacterial effect of these growth factors has been reported.

To better efficacy and comfortable utilization of platelet, it is feasible to form the platelet gel and then apply on wound sites.

This study is a double blind randomized controlled trial to evaluate the positive effects of umbilical cord blood-derived platelet gel in 244 patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
In this study all qualified patients (based on the inclusion and exclusion criteria) were randomly allocated into three study groups by a Stratified Permuted Block randomization method: group A received platelet rich plasma gel, group B (placebo) received platelet poor plasma gel, and group C received lubricant gel.

All of the patients underwent a standard long protocol for knee osteoarthritis. All patients with diabetic foot ulcer are selected.On average,in each instance, the amount of platelets in the peripheral bloodis4 to6 times the baseline level.

Group A (interventional): application of 20-30mL of gel from platelet rich plasma (PRP) Group B (placebo): application of 20-30mL of gel from platelet poor plasma (PRP) Group C (control): application of 20-30 mL of lubricant gel (used typically for sonography)

ELIGIBILITY:
Inclusion Criteria:

* History of at least 4 weeks hospitalization
* Uncontrolled diabetes
* ejection fraction > 30%

Exclusion Criteria:

* mechanical origin for wound
* history of infectious, systemic diseases, Immune deficiency and coagulation disorders

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
pain | 3 months
  Evaluation the pain reduction by VAS measurement in patients with peripheral artery Disease.
ABI | 3 months
  Evaluation the Ankle Brakial Index (ABI) in patients 3 months after PG utilization.

SECONDARY OUTCOMES:
Quality of life | 3months
  Evaluation the quality of life by SF36 measurement in patients with PAD.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of regenerative medicine department &cell therapy center of Royan Institute; Behnam Molavi, MD, Study Director — Department of vascular & Trauma Surgery of Sina Hospital; Seyedeh Esmat Hosseini, Bs, Principal Investigator — Department of Regenerative Medicine & cell therapy of Royan Institute; Alireza Goodarzi, MSc, Principal Investigator — Department of Regenerative Medicine of Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org